CLINICAL TRIAL: NCT00992836
Title: A Phase II Study to Assess the Safety and Immunogenicity of an Inactivated Swine-Origin H1N1 Influenza Vaccine in HIV-1 Perinatally Infected Children and Youth
Brief Title: Safety of and Immune Response to an H1N1 Influenza Virus Vaccine in HIV Infected Children and Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P1088; 10840 (Registry Identifier: DAIDS ES Registry Number); IMPAACT P1088
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2014-12

CONDITIONS: HIV Infections; H1N1 Influenza Virus
Keywords: Influenza A Virus, H1N1 Subtype; Vaccine; Children; Adolescents; HIV-Infected; Perinatal HIV Infection; Treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Influenza A (H1N1) 2009 monovalent vaccine (Experimental): All participants received two doses of the H1N1 influenza virus vaccine, administered 21 days apart.
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine

INTERVENTIONS:
Biological: Influenza A (H1N1) 2009 monovalent vaccine — Two doses of vaccine, delivered 21 days apart, with each dose consisting of two 15-microgram intramuscular injections

SUMMARY:
Children and people infected with HIV are particularly susceptible to influenza infections. This study testED the safety and effectiveness of a vaccine for the new H1N1 influenza virus in children and youth infected with HIV.

DETAILED DESCRIPTION:
The new H1N1 influenza virus seen in 2009 has been designated a pandemic by the World Health Organization, due to the sustained community outbreaks seen in the United States and Mexico. Based on preliminary data, it appears children and young adults were particularly at risk of the H1N1 virus. People infected with HIV were also more susceptible to severe influenza infections than those who are uninfected. Children with HIV infection, then, have a compounded risk of H1N1 infection. Higher doses of influenza vaccines are associated with the development of higher levels of serum antibodies, which are needed to resist infection. Higher vaccine doses can be used to improve vaccine effectiveness in at-risk populations. This study tested the safety and immune response of HIV infected children and youth to a high dose of a vaccine for the new H1N1 influenza virus.

Participation in this study lasted 7 months and had two steps. The first step involved receiving the first dose of H1N1 virus vaccine, and the second step, occurring 21 days later, involved receiving the second dose of vaccine. Each dose of vaccine was delivered via two intramuscular shots (four total injections). After receiving each dose of the vaccine, participants were given a diary to record any symptoms or reactions. Participants were stratified into three groups by age, including 4 to 9 years, 9 to 18 years, and 18 to 25 years.

Participants completed five scheduled visits, taking place at screening, study entry, Days 21 and 31, and after 7 months. Measurements taken on these visits included a medical history, physical and neurological exams, a blood draw, and, when applicable, a pregnancy test. In addition to these visits, participants received up to three additional phone calls or visits occurring 2 and 10 days after the first dose of vaccine and 2 days after the second dose of vaccine to check for reactions to the vaccine.

ELIGIBILITY:
Inclusion Criteria for Step I:

* HIV infected
* HIV-1 was perinatally acquired, in the opinion of the investigator
* Participants receiving antiretrovirals (ARVs) must have been receiving a stable regimen for 90 days prior to entry with no intention to modify their regimen within 60 days following study entry
* Participants not receiving ARVs at entry must not have received ARVs within 90 days prior to entry and must NOT plan to initiate ARVs within 60 days following study entry
* Ability to complete all study immunizations and evaluations, in the opinion of the investigator
* Agrees to use contraception, if necessary
* Documented platelet count of more than 50,000 per mm3 and an absolute neutrophil count (ANC) of more than 500 per mm3 within the 30 days prior to study entry
* Youth of legal age (from 18 to 25 years of age), parent or legal guardian, or participants who are emancipated minors must provide informed consent

Inclusion Criteria for Step II:

* Received the first dose of Influenza A (H1N1) 2009 monovalent vaccine at least 21 days ago
* Documented platelet count of more than 50,000 per mm3 and an ANC of more than 500 per mm3 within the 30 days prior to Step II entry
* If a woman became pregnant after Dose #1, she must be at more than 14 weeks of gestation and have her obstetrician's permission to receive the vaccine

Exclusion Criteria for Step I:

* Pregnancy
* Known allergy to egg protein (egg or egg product) or other components in the vaccines (these may include, but are not limited to: neomycin and polymyxin)
* History, in the opinion of the site investigator, of severe reactions following previous immunization with seasonal influenza vaccines that would contraindicate receipt of any influenza vaccine.
* History of probable or proven pandemic 2009 Influenza A (H1N1) infection prior to study entry
* Has received any live licensed vaccine within 4 weeks or inactivated licensed vaccine within 2 weeks prior to study entry
* Has received a nonlicensed agent (vaccine, drug, biologic, device, blood product, or medication) within 4 weeks prior to study entry or expects to receive another nonlicensed agent during the course of the study
* Has an acute illness or a documented temperature greater than or equal to 100.0 degrees Fahrenheit within 24 hours prior to study entry
* Use of anti-cancer chemotherapy or radiation therapy within the 36 months preceding study entry or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection)
* Has an active neoplastic disease
* Long-term use of glucocorticoids, including oral or parenteral prednisone or equivalent (at least 2 mg/kg per day or at least 20 mg total dose) for more than 2 weeks in the past 6 months or high-dose inhaled steroids (more than 800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. Nasal and topical steroids are allowed.
* Has received immunoglobulin or other blood products within the 3 months prior to study entry
* History of Guillain-Barre syndrome in the subject or subject's family, including parents, siblings, half-siblings, and children
* Onset of a neurological disorder including (but not limited to) absent ankle and patellar deep tendon reflexes in both legs (all four absent) within the past 6 months
* Disproportionate loss of strength in lower extremity or extremities compared to the upper extremities within the past 6 months
* Has any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Exclusion Criteria for Step II:

* Has received a nonlicensed agent (vaccine, drug, biologic, device, blood product, or medication), other than from participation in this study, since Dose #1 or expects to receive another nonlicensed agent before the end of the study
* Use of anti-cancer chemotherapy or radiation therapy since Dose #1, new diagnosis of an active malignancy, or is immunosuppressed as a result of an underlying illness (other than HIV-1 infection) or treatment.
* Use of glucocorticoids, including oral or parenteral steroids (at least 2 mg/kg per day or at least 20 mg total dose) for more than 2 weeks since vaccine Dose #1 or high-dose inhaled steroids (more than 800 mcg/day of beclomethasone dipropionate or equivalent) since Dose #1 (nasal and topical steroids are allowed)
* Has received immunoglobulin or other blood products since Dose #1
* Any Grade 3 toxicity or adverse event (AE) experienced by a participant, unless the investigator has received protocol team approval
* Any Grade 4 toxicity or AE (other than injection site reaction or fever) that is definitely, probably or possibly related to study vaccine
* Any Grade 4 injection site reactions or fever experienced by a participant, unless the investigator has received protocol team approval
* Any Grade 4 AEs that are definitely not or probably not related to study vaccine, unless the investigator has received protocol team approval
* New occurrence or new awareness of Guillain-Barre syndrome in the participant or participant's family (parents, siblings, half-siblings, or children) since Dose #1
* New onset of a neurological disorder including (but not limited to) absent ankle and patellar deep tendon reflexes in both legs (all four absent) since Dose #1
* Disproportionate loss of strength in lower extremity or extremities compared to the upper extremities (not thought to be related to pregnancy) since Dose #1
* Documented infection with 2009 Influenza A (H1N1) since Dose #1
* Refusal of further vaccination by participant, parent, or guardian
* Development of any new disease that the investigator judges to be clinically significant or clinically significant findings since Dose #1 that, in the investigator's opinion, would compromise the safety of the subject
* Withdrawal of consent. Consent may be withdrawn at any time and for any reason, without penalty.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pat Flynn, MD, Study Chair — St. Jude Children's Research Hospital
Locations (37):
- United States (35):
  - UAB Pediatric Infectious Diseases CRS, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Harbor UCLA Medical Ctr. NICHD CRS, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Puerto Rico (2):
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Gelinck LB, van den Bemt BJ, Marijt WA, van der Bijl AE, Visser LG, Cats HA, Rimmelzwaan GF, Kroon FP. Intradermal influenza vaccination in immunocompromized patients is immunogenic and feasible. Vaccine. 2009 Apr 21;27(18):2469-74. doi: 10.1016/j.vaccine.2009.02.053. Epub 2009 Feb 24. PMID 19368788
- [Result] Flynn P, Nachman S, Spector SA, Cunningham CK, Weinberg A, Pass R, Muresan P, Levy W, Siberry G, Handelsman E for the IMPAACT P1088 and P1089 Teams: Safety and Immunogenicity of 2009 H1N1 Influenza Immunization in HIV-1 Perinatally Infected Children and Youth. Presented at the IDSA conference, October 2010.
- [Result] Flynn PM, Nachman S, Spector SA, Cunningham CK, Weinberg A, Pass R, Muresan P, Levy W, Petzold E, Heckman B, Siberry G, Handelsman E for the IMPAACT P1088 and P1089 Teams. 2009 Influenza A (H1N1) Immunization in HIV-1 Perinatally Infected Children and Youth. Presented at the Retroviruses Conference, Feb 2010.
- [Derived] Curtis DJ, Muresan P, Nachman S, Fenton T, Richardson KM, Dominguez T, Flynn PM, Spector SA, Cunningham CK, Bloom A, Weinberg A. Characterization of functional antibody and memory B-cell responses to pH1N1 monovalent vaccine in HIV-infected children and youth. PLoS One. 2015 Mar 18;10(3):e0118567. doi: 10.1371/journal.pone.0118567. eCollection 2015. PMID 25785995
- [Derived] Flynn PM, Nachman S, Muresan P, Fenton T, Spector SA, Cunningham CK, Pass R, Yogev R, Burchett S, Heckman B, Bloom A, Utech LJ, Anthony P, Petzold E, Levy W, Siberry GK, Ebiasah R, Miller J, Handelsman E, Weinberg A; IMPAACT P1088 Team. Safety and immunogenicity of 2009 pandemic H1N1 influenza vaccination in perinatally HIV-1-infected children, adolescents, and young adults. J Infect Dis. 2012 Aug 1;206(3):421-30. doi: 10.1093/infdis/jis360. Epub 2012 May 21. PMID 22615311
- See also: Click here for information on the IMPAACT group and for the package insert on the H1N1 vaccine. — http://www.impaactgroup.org/
- See also: Click here for the table used for grading toxicities: DAIDS Grading Severity of AEs, V1.0, Dec04. — http://rsc.tech-res.com/safetyandpharmacovigilance/gradingtables.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 37 sites between October 14, 2009 and November 12, 2009. Participants were stratified by age in three groups: >=4 to < 9 years old, >=9 to < 18 years old and >=18 to <25 years old.
Pre-assignment Details: One study participant was inadvertently enrolled with acute illness, was not given any vaccination and was immediately taken off study. A second study participant received the first vaccination but it was discovered that he/she was not compliant with the ARV regimen and was taken off study before receiving the second dose of vaccine.
Groups:
- All Study Participants: Participants received two doses of the H1N1 influenza virus vaccine, administered 21 days apart. Each dose consisted of two 15-microgram intramuscular injections.
Period: Overall Study
Arm/Group | All Study Participants
Started | 155
Received Both Study Vaccinations | 150
Completed | 150
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 79
Region of Enrollment [Number; unit: participants]
  United States | 147
  Puerto Rico | 8
Age Strata [Number; unit: Participants] — Study participants were stratified by age into three groups.
  Participants
    >=4 to < 9 years old | 54
    >=9 to < 18 years old | 51
    >=18 to < 25 years old | 50
CD4 Cells Count [Mean (Standard Deviation); unit: cells / mm^3] — This measures the number of CD4 cells.
  cells / mm^3 | 568 (242)
Percentage of CD4 Cells [Mean (Standard Deviation); unit: percentage] — This measures the percentage of CD4 cells.
  percentage | 29 (11)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Had at Least One Adverse Event (AE)
Description: Shows the number of participants who had at least one adverse event (AE) in each category. The AEs include: abnormal laboratory values, signs and symptoms, or diagnoses; solicited local AEs; and solicited systemic AEs.
  Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Time Frame: Measured up to 7 months after vaccination
Measure: Number; unit: participants
Groups:
- All Study Participants: All 155 study participants are included in this analysis.
Arm/Group | All Study Participants
Number analyzed (Participants) | 155
participants
  Overall (New AEs after start of treatment) | 113
  Grade 4 AEs (New, after start of treatment) | 0
  Grade 3 AEs (New, after start of treatment) | 7
  Grade 2 local and systemic AEs to injection | 6

2. Primary Outcome: The Number of Participants Who Had at Least One AE Attributed to the Study Vaccine
Description: Shows the number of participants who experienced any events that were thought to be at least possibly related to study treatment. Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Time Frame: Measured up to 7 months after vaccination
Population: The 154 study participants who received at last one vaccination are included in this analysis.
Measure: Number; unit: participants
Groups:
- Vaccinated Study Participants: The 154 study participants who received at last one vaccination are included in this analysis.
Arm/Group | Vaccinated Study Participants
Number analyzed (Participants) | 154
participants | 7

3. Primary Outcome: Withholding of Second Vaccine Dose Due to Adverse Reactions Attributed to First Dose
Time Frame: Measured at Day 21
Population: The 154 study participants who received at last one vaccination are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Vaccinated Study Participants
Number analyzed (Participants) | 154
participants | 0

4. Primary Outcome: Percent of Participants With a Hemagglutinin Inhibition (HAI) Titer of >=40
Description: Antibodies to Influenza A (H1N1) 2009 were measured using an HAI assay. The potential titer read-outs from the assay used were <10 (considered undetectable), 10, 20, 40, 60, 80, 160, 320, 640 and >=1280. Seroprotection was defined as having a titer of >=40 following vaccination.
Time Frame: Measured at 21 days after first dose and 10 days after second dose
Population: The HAI titers following the first vaccination were summarized for the eligible study participants who received at least one vaccine and had nonmissing HAI data, and the titers following the second vaccination for the eligible study participants who received both doses of vaccine and had nonmissing HAI data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall: The total N for these analyses were 140 and 142, for the analysis of antibody titers after the first and second vaccinations, respectively.
Arm/Group | Overall
Number analyzed (Participants) | 142
percentage of participants
  Post dose 1 (N=140) | 72.1 [63.9 to 79.4]
  Post dose 2 (N=142) | 82.4 [75.1 to 88.3]

5. Secondary Outcome: Percent of Participants With an HAI Titer >=40 at Long-term Follow-up
Time Frame: Measured at 6 months after second dose
Population: The HAI titers were summarized for the eligible study participants who received both doses of vaccine and had nonmissing HAI data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall: The total N for this analysis was 138, those who received both vaccinations and had nonmissing data.
Arm/Group | Overall
Number analyzed (Participants) | 138
percentage of participants | 57.2 [48.5 to 65.6]

6. Secondary Outcome: Geometric Mean Antibody Titers (GMT) HAI
Description: Presents the value of the geometric mean titer at each time point.
Time Frame: Measured after first and second doses and 6 months after second dose
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Overall: The total N for these analyses were 140, 142 and 138, for the analysis of antibody titers after the first and second vaccinations and after 6 months after the second vaccination, respectively.
Arm/Group | Overall
Number analyzed (Participants) | 142
titers
  At 21 days after the first vaccination (N=140) | 85 [65 to 111]
  At 10 days after the second vaccination (N=142) | 127 [101 to 159]
  At 6 months after the second vaccination (N=138) | 33 [27 to 40]

7. Secondary Outcome: Cell-mediated Immune Responses, Measured by B-cell and T-cell Enzyme-linked Immunosorbent Spot (ELISPOT) Assay Values
Description: The median and interquartile range (IQR) of B-Cell ELISPOT-measured IgG antibody-secreting cells (ASC)/10^6 peripheral blood mononucleated cell (PBMC) and the median and interquartile range (IQR) of T-Cell ELISPOT-measured pH1N1 IFNgamma spot-forming cells (SFC)/10^6 PBMC.
Time Frame: Measured at entry, 21 days after first dose, and 10 days after second dose
Population: The participants who had received all doses of vaccine up to that timepoint and had sufficient samples for testing.
Measure: Median (Inter-Quartile Range); unit: ASC or SFC/10^6 PBMC
Groups:
- Overall: The total N for this analysis was 68, those who received the vaccinations and had enough samples for testing.
Arm/Group | Overall
Number analyzed (Participants) | 68
ASC or SFC/10^6 PBMC
  IgG ASC/10^6 PBMC, Week 0 (N=46) | 6 [2 to 16]
  IgG ASC/10^6 PBMC, Post Dose 1 (N=40) | 13 [4 to 40]
  IgG ASC/10^6 PBMC, Post Dose 2 (N=40) | 12 [5 to 25]
  pH1N1 IFNgamma SFC/10^6 PBMC, Week 0 (N=68) | 317 [117 to 673]
  pH1N1 IFNgamma SFC/10^6 PBMC, Post Dose 1 (N=68) | 363 [123 to 622]
  pH1N1 IFNgamma SFC/10^6 PBMC, Post Dose 2 (N=65) | 261 [78 to 525]

8. Secondary Outcome: HAI Titers Against Seasonal Influenza Viruses Containing Trivalent Influenza Vaccine (TIV)
Description: Presents the value of the median titer as well as the interquartile range at study entry. Antibodies to seasonal Influenza vaccine were measured using an HAI assay. The potential titer read-outs from the assay used were <10 (considered undetectable), 10, 20, 40, 60, 80, 160, 320, 640, and >=1280.
Time Frame: Measured at entry, 21 days after first dose, and 10 days and 6 months after second dose
Population: The participants who had received all doses of vaccine up to that timepoint and had sufficient samples for testing.
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | Influenza A (H1N1) 2009 Monovalent Vaccine
Number analyzed (Participants) | 123
titer
  Week 0 (N=123) | 40 [20 to 80]
  Post Dose 1 (N=121) | 40 [20 to 80]
  Post Dose 2 (N=121) | 40 [20 to 80]
  6 months Post Dose 2 (N=122) | 40 [20 to 80]

9. Secondary Outcome: Cell-mediated Immune Responses to Influenza Viruses Contained in TIV and Other Antigens
Description: The TIV assay was not performed due to lack of available cells after completion of other planned assays.
  The median and interquartile range (IQR) of T-Cell ELISPOT-measured pH1N1 Granzyme B spot-forming cells (SFC)/10^6 peripheral blood mononucleated cell (PBMC).
  The median and interquartile range (IQR) of T-Cell ELISPOT-measured PHA INFgamma spot-forming cells (SFC)/10^6 PBMC.
  The median and interquartile range (IQR) of T-Cell ELISPOT-measured PHA Granzyme B spot-forming cells (SFC)/10^6 PBMC.
Time Frame: Measured at entry, 21 days after first dose, and 10 days after second dose
Population: The participants who had received all doses of vaccine up to that timepoint and had sufficient samples for testing.
Measure: Median (Inter-Quartile Range); unit: SFC/10^6 PBMC
Arm/Group | Overall
Number analyzed (Participants) | 68
SFC/10^6 PBMC
  pH1N1 Granzyme B SFC/10^6 PBMC, Week 0 (N=64) | 35 [0 to 220]
  pH1N1 Granzyme B SFC/10^6 PBMC, Week 3 (N=62) | 26 [0 to 170]
  pH1N1 Granzyme B SFC/10^6 PBMC, Week 5 (N=61) | 30 [0 to 220]
  PHA INFgamma SFC/10^6 PBMC, Week 0 (N=68) | 699 [307 to 1010]
  PHA INFgamma SFC/10^6 PBMC, Week 3 (N=68) | 637 [261 to 965]
  PHA INFgamma SFC/10^6 PBMC, Week 5 (N=65) | 624 [263 to 1000]
  PHA Granzyme B SFC/10^6 PBMC, Week 0 (N=64) | 3250 [390 to 7465]
  PHA Granzyme B SFC/10^6 PBMC, Week 3 (N=62) | 3340 [510 to 7520]
  PHA Granzyme B SFC/10^6 PBMC, Week 5 (N=60) | 2045 [300 to 7825]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of enrollment in the study until 6 months after second vaccination.
Description: Include Adverse Events (AEs) of All Grades, Including Abnormal Laboratory Values, Signs and Symptoms, or Diagnoses; Solicited Local AEs and Systemic AEs. Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 6/155
Other Adverse Events (participants affected / at risk) | 113/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=155)
Neutropenia (Blood and lymphatic system disorders) | 1
Gait disturbance (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=155)
Ear pain (Ear and labyrinth disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 18
Adverse event (General disorders) | 20
Fatigue (General disorders) | 11
Pyrexia (General disorders) | 19
Otitis media (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 9
Neutrophil count decreased (Investigations) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 51
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 35
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No